CLINICAL TRIAL: NCT00579306
Title: Levels of Inflammatory Markers in the Treatment of Stroke
Brief Title: Levels of Inflammatory Markers in the Treatment of Stroke-An SPS3 Ancillary Study
Acronym: LIMITS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Mitchell S Elkind, Associate Professor of Neurology and Epidemiology (in the Sergievsy Center), Columbia University
Other Study IDs: AAAB1202; R01NS050724 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Hypertension; Stroke
Keywords: hypertension; stroke; cerebrovascular accident
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum (ancillary study)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPS3 patient cohort: All SPS3 patients who participate in Baseline and 1-Year F/U blood draw

SUMMARY:
The goals of this trial are to determine the prognostic significance of an elevated level of inflammatory blood markers in people who have experienced small subcortical strokes and who are enrolled in the Secondary Prevention of Small Subcortical Strokes (SPS3) trial.

DETAILED DESCRIPTION:
Inflammation is increasingly recognized as playing a central role in atherosclerosis and coronary artery disease. And, peripheral blood markers of inflammation have been associated with incident and recurrent cardiac events. The relationship of these risk markers-which have the potential to be modified-to prognosis after ischemic stroke is less clear.

The Levels of Inflammatory Markers in the Treatment of Stroke (LIMITS) study will address questions about the role of inflammatory markers in secondary stroke prevention in a cost-effective manner using the well-established framework of the Secondary Prevention of Small Subcortical Strokes (SPS3) trial. The SPS3 trial is an ongoing Phase 3, multicenter secondary stroke prevention trial that focuses on preventing stroke recurrence in people with small vessel ischemic stroke, or lacunes.

The overall purpose of the LIMITS study is to determine if serum levels of inflammatory markers-such as hsCRP, serum amyloid A (SAA), CD40 ligand (CD40L), and monocyte chemoattractant protein-1 (MCP-1)-predict recurrent stroke and other vascular events among people with a history of small artery ischemic stroke. The project will also determine if these markers predict which people will respond best to dual antiplatelet therapy with clopidogrel and aspirin.

The specific aims of LIMITS are to determine if hsCRP, SAA, CD40L, and MCP-1 levels are independent risk factors for recurrent ischemic stroke, and for recurrent ischemic stroke, myocardial infarction, and death in participants in the SPS3 trial after adjusting for demographic and traditional stroke risk factors, and other treatments, using a prospective cohort of people with small subcortical strokes from the SPS3 trial. LIMITS also aims to compare the efficacy of dual versus single antiplatelet therapy among participant groups with and without elevated baseline inflammatory marker levels for the outcome of a.) recurrent stroke, and b.) recurrent ischemic stroke, myocardial infarction, or death.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be randomized within 6 months of qualifying small subcortical stroke (S3) or subcortical TIA
* One of the following lacunar syndromes: PMH; pure sensory stroke; sensorimotor stroke; ataxic hemiparesis; dysarthria; hemiballism; PMH with facial sparing, horizontal gaze palsy, contralateral III palsy, contralateral VI palsy; Ataxia with contralateral III palsy; pure dysarthria
* Absence of cortical dysfunction (aphasia, apraxia, agnosia)
* No ipsilateral cervical carotid stenosis (>= 50%) if S3 is hemispheric
* No major-risk cardioembolic sources requiring anti-coagulation
* MRI evidence of S3 that is >=2.0 cm in diameter if DWI/bright lesion on FLAIR/T2 or <=1.5cm hypointense lesion on FLAIR/T1, corresponding to the qualifying event (required for all brainstem events) OR multiple S3 in cerebral hemispheres of <=1.5cm hypointense lesions on FLAIR/T1 AND absence of cortical stroke and large subcortical stroke.

Exclusion Criteria:

* Disabling stroke (Ranking Scale >= 4)
* Prior hemorrhagic stroke
* Age <30 years
* High risk of bleeding (recurrent GI or GU bleeding, active peptic ulcer disease, etc)
* Need for long-term use of anticoagulants or other antiplatelet agents.
* Prior cortical or retinal stroke / TIA
* Prior ipsilateral carotid endarterectomy if hemispheric S3
* Impaired renal function: GFR<40 cc/min
* Intolerance/contraindication to aspirin or clopidogrel
* Adjusted Folstein MMSE <24
* Medical contraindication to MRI
* Pregnancy or child-bearing potential without contraception
* Other specific causes of stroke (e.g. dissection, vasculitis, drug abuse)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a symptomatic small vessel stroke within prior 6 month and enrolled in SPS3
Sampling Method: Probability Sample
Enrollment: 1244 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with recurrent stroke | Up to 5 years
  Participants with recurrence of any stroke during follow-up, including ischemic (an acute localized ischemic lesion in the brain not attributable to central nervous system infection, tumor, demyelinating, or degenerative neurologic diseases due to an occlusive vascular disorder) and hemorrhagic (acute extravasation of blood into the parenchyma of the central nervous system or subarachnoid space).

SECONDARY OUTCOMES:
Percentage of participants developing major cognitive decline | Up to 5 years
  Documentation of a major cognitive decline during follow-up. This is a clinical decline in cognitive function manifested by functional deterioration/behavioral changes that are not associated with a clinical stroke event.
  Criteria: Both A and B must be met:
  A) A drop in the Cognitive Abilities Screening Instrument (CASI) score of > 10 points since study entry and sustained on repeat testing in approximately one month B) Associated behavioral changes and/or function

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Elkind, MD, MS, FAAN, Principal Investigator — Columbia University; Oscar Benavente, MD, Principal Investigator — UTHSC San Antonio (SPS3 Principal Investigator); Robert Hart, MD, Principal Investigator — UTHSC San Antonio (SPS3 Principal Investigator)
Locations (45):
- United States (30):
  - University of South Alabama, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arizona Collage of Medicine, Tucson, Arizona
  - University of California, San Diego Medical Center, La Jolla, California
  - Sutter Neuroscience Institute, Sacramento, California
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - University of Miami, Miami, Florida
  - Mercy Medical Center, Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Boston University Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Cooper University Hospital,, Camden, New Jersey
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Helen Hayes Hospital, West Haverstraw, New York
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Case Western Reserve University,Case Western Neurological Unit, 11100 Euclid Avenue, Lakeside 5508, Cleveland, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas South Western Medical Center, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Dalhousie University Center for Clinical Research, Halifax, Nova Scotia
  - Hospital Charles LeMoyne Centre de recherché, Greenfield Park, Quebec
  - McGill University Health Center, Montreal, Quebec
- Chile (2):
  - Pontificia Universidad Catolica de Chile, Santiago
  - Hospital Naval Almirante Nef, Viña del Mar
- Hospital-Clinica Kennedy, Guayaquil, Ecuador
- Mexico (2):
  - Universidad Autonoma de Guadalajara, Guadalajara, Jalisco
  - Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico City
- Hospital Nacional Alberto Sabogal, Lima, Peru
- Spain (6):
  - Hospital Clinico Universitario de Santiago de Compostela, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital del Sagrat Cor, Barcelona
  - Hospital Dr. Josep Trueta, Barcelona
  - Hospital Germans Trias i Pujol,, Barcelona
  - Hospital Universitario de Bellvitge, Spain, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided